CLINICAL TRIAL: NCT03818412
Title: Circulating Tumor DNA Detection in Soft Tissue Sarcoma (DNA-TSAR)
Brief Title: Circulating Tumor DNA in Soft Tissue Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DNA-TSAR
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Soft Tissue Sarcoma
Keywords: Circulating tumor DNA
MeSH Terms: conditions — Sarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soft Tissue Sarcoma (Experimental): A sample of archival tumor tissue will be collected.
  Blood samples (about 20-30 mL or 1-2 tablespoons each sample) will be taken:
  * Prior to planned radiation treatment
  * 2-4 weeks after cancer surgery
  * Every 12 weeks after surgery for up to 2 years
  Interventions: Procedure: Archival tumor tissue collection and blood draws

INTERVENTIONS:
Procedure: Archival tumor tissue collection and blood draws — Archival tumor tissue will be collected for testing of circulating tumor DNA. Blood draws will be taken for testing of circulating tumor DNA.

SUMMARY:
This research study will collect blood and tumor tissue samples from patients with soft tissue sarcoma to look at circulating tumor deoxyribonucleic acid (DNA). When tumor cells are damaged or die, DNA from the tumor cells are released into the blood stream as the cells break down. This is called circulating tumor DNA. Circulating tumor DNA is an important biomarker that may be used in cancer detection, prediction of treatment response, and disease monitoring.

DETAILED DESCRIPTION:
Researchers are continually looking for ways to understand the biology of cancer such as sarcoma, and ways to improve cancer care and patient outcome.

Research has shown that changes in some genes and/or proteins, called biomarkers, may be important indicators for certain cancers and response to treatments. Genes are molecules made up of ribonucleic acid (RNA) and deoxyribonucleic acid (DNA). DNA contain instructions for the development and functioning of the cells in the body and are passed down from parent to child. RNA is involved with producing proteins in the body. Further research is needed to better understand the changes found in cancer cells and what this means for certain treatments.

Circulating tumor DNA is an important biomarker that may be used in cancer detection, prediction of treatment response and disease monitoring. When tumor cells are damaged or die, DNA from the tumor cells are released into the blood stream as the cells break down. This is called circulating tumor DNA. Researchers are looking for better ways to detect circulating tumor DNA so that it can be studied.

The purpose of this study is to determine how feasible it is to detect circulating tumor DNA in blood samples of soft tissue sarcoma patients and whether there is a connection between circulating tumor DNA and the likelihood of patients' disease coming back after they receive treatment. To do this, blood and tumor tissue samples will be collected from participants and will undergo DNA testing (reading the contents of their DNA, called sequencing). The results of the DNA testing in the blood samples will be compared with the results from DNA testing that will also be done on tumor tissue. The results will also be compared with participant's response to their treatment, recurrence, and/or long term survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed high-risk extremity or retroperitoneal liposarcoma, leiomyosarcoma and undifferentiated pleomorphic sarcoma.
* Patients must have archival tissue from the diagnostic biopsy available.
* Deemed appropriate for preoperative or postoperative radiotherapy and curative surgery following patient assessment by radiation oncologist and surgical oncologist.
* Age 18 years or older.
* Eastern Cooperative Group (ECOG) performance status ≤ 2
* Ability to understand and willing to sign a written informed consent document and comply with study requirements.

Exclusion Criteria:

* Patients with benign histology
* Patients with prior malignancy within previous 5 years or concurrent malignancy other than adequately treated basal cell carcinoma of skin or carcinoma in-situ of cervix.
* Patients with planned neo-adjuvant chemotherapy.
* Patients with regional nodal disease or unequivocal metastases
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2024-12-17 (Estimated); Study Completion 2025-01-17 (Estimated)

PRIMARY OUTCOMES:
Number of patients with demonstrable circulating tumor DNA (ctDNA) quantification | 5 years
  Duration from time of study trial until end

SECONDARY OUTCOMES:
Number of patients with demonstrable ctDNA quantification with no pre-op tumor burden, necrosis at surgery, or disease recurrence | 5 years
  Duration from time of study trial until end

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni Razak, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada